CLINICAL TRIAL: NCT01951248
Title: Central and Peripheral 24-h Blood Pressure Measurements in Patients With Chronic Renal Failure and Obstructive Sleep Apnea Before and After Treatment With CPAP
Brief Title: Central and Peripheral 24-h Blood Pressure Before and After 3 Month of CPAP Treatment in Obstructive Sleep Apnea
Acronym: NOSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Professor, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGH-3-2013; M-2013-285-13 (Other: The Regional Commitww of Health Research Ethics)
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Kidney Disease; Obstructive Sleep Apnea
Keywords: chronic kidney disease; obstructive sleep apnea; 24-h blood pressure; central blood pressure; peripheral blood pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP treatment (Experimental): Patients with chronic kidney disease and moderate to severe obstructive sleep apnea is treated 3 months with CPAP treatment
  Interventions: Device: CPAP - continuous airway pressure

INTERVENTIONS:
Device: CPAP - continuous airway pressure — 3 months of treatment with CPAP treatment
  Other Names: S9 AutoSet from ResMed/Maribo Medico; or; REMstar Auto A-Flex from Phillips/Respirsonics

SUMMARY:
The purpose of this study is to investigate the effect of 3 months of continuous positive airway pressure (CPAP) treatment of obstructive sleep apnea (OSA) in moderate to severe cases in patients with chronic kidney disease. The effect is evaluated on blood pressure levels, particularly nocturnal blood pressure, both central and peripheral, and renal function, including the kidneys treatment of salt and water.

Hypothesis:

1. Central 24-h blood pressure measuring is a reveals fluctuations in blood pressure during the day more accurately than peripheral 24-h blood pressure measuring because the measurement is painless and does not interfere with the patient activities during the daytime or nighttime sleep.
2. Central blood pressure is elevated in patients with OSA and falls during treatment with CPAP.
3. The renal tubular function relating to the treatment of water and sodium is abnormal in patients with OSA with increased tubular absorption of water via the U-aquaporin 2 (u-AQP2) and of sodium by epithelial sodium channel (ENAC) and is normalized during treatment with CPAP.

4 Quality of life is improved during treatment with CPAP.

DETAILED DESCRIPTION:
Approximately 30 patients with chronic kidney disease and obstructive sleep apnea in moderate to severe degree is examined with central and peripheral 24-h blood pressure monitoring, 1 night home polygraphy to determine the degree of sleep apnea, blood and urine samples to determine levels of u-AQP2, u-ENAC, plasma renin concentration (PRC), s-angiotensin II (p-angII), p-aldosterone, p-vasopressin (p-avp) and p-endothelin, before the start treatment with CPAP for sleep apnea.

After 3 month of treatment all the above described is repeated to determine effects of CPAP treatment on blood pressure levels during the day, changes i apnea hypopnea index (AHI) and the kidneys treatment of salt and water.

ELIGIBILITY:
Inclusion Criteria:

* renal insufficiency (CKD stage III + IV), estimated glomerular filtration rate (eGFR) 15-59 ml/min/1.73 m2
* Obstructive sleep apnea, AHI> 15 (moderate to severe)
* both men and women
* 18-80 years

Exclusion Criteria:

* lack of desire to participate
* malignant disease
* Abuse of drugs or alcohol
* pregnant and lactating
* incompensated heart failure
* atrial fibrillation
* liver disease (alanine aminotransferase> 200)
* Severe chronic obstructive lung disease (Forced expiratory volume in 1 second <50% predicted)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
decrease in systolic night time blood pressure | 3 months
  The difference in systolic blood pressure at night by 24-h blood pressure at baseline and 3 months of treatment of OSA with CPAP in patients with chronic renal insufficiency.

SECONDARY OUTCOMES:
difference in systolic blood pressure at night by central blood pressure monitoring | 3 months
  The difference in systolic blood pressure at night by central 24-h blood pressure monitoring before and after 3 months of treatment of OSA with CPAP in patients with chronic renal insufficiency
systolic and diastolic blood pressure throughout the day | 3 months
  The difference in systolic blood pressure and diastolic blood pressure throughout the day, in the daytime and in night time between measurements with peripheral 24-h blood pressure and central 24-h blood pressure before and after 3 months of treatment with CPAP.
correlation between blood pressure, OSA and kidney function | 3 months
  The correlation between the treatment effect on blood pressure levels on the one hand and the severity of OSA prior to initiation of treatment and renal function measured by estimates glomerular filtration rate, on the other
U-AQP2 and u-ENaCɣ in day urine. PRC, p-AngII, p-Aldo. P-AVP and p-endothelial. | 3 months
  U-AQP2 and u-ENaCɣ in day urine. PRC, p-AngII, p-Aldo. P-AVP and p-endothelial. Difference in these before and after 3 months of treatment
quality af life | 3 months
  difference in the quality of life before and after 3 months of CPAP treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medicinsk Forskning, Holstebro, Holstebro, Denmark